CLINICAL TRIAL: NCT02612077
Title: A Cohort Survey of Patients With Metastatic Colorectal Cancer Starting a Chemotherapy in Combination With Avastin®
Brief Title: Observation of Patients With Metastatic Colorectal Cancer Starting Chemotherapy Combined With Bevacizumab (Avastin)
Acronym: CONCERT
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21696
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational Chemotherapy/Bevacizumab: Observed patients receiving chemotherapy with concomitant bevacizumab
  Interventions: Other: Observational Chemotherapy; Drug: Concomitant Bevacizumab

INTERVENTIONS:
Other: Observational Chemotherapy — No intervention - Observational standard practice chemotherapy
Drug: Concomitant Bevacizumab — No intervention - Observational concomitant bevacizumab
  Other Names: Avastin

SUMMARY:
This is a longitudinal, multicenter, prospective, pharmacoepidemiological study to evaluate progression free survival (PFS) in a real-life setting in participants with metastatic colorectal cancer (mCRC) starting chemotherapy combined with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Having colon or rectal metastatic adenocarcinoma, for which the physician decided during the inclusion visit to start a treatment with bevacizumab combined with a 1st, 2nd or 3rd line chemotherapy
* Having received oral and written information about the survey and not objecting to having his/her data computerized

Exclusion Criteria:

- Participating in a clinical trial assessing an anticancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer (mCRC) starting chemotherapy combined with bevacizumab.
Sampling Method: Non-Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2008-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuilly-sur-Seine, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational Chemotherapy/Bevacizumab
Started | 765
Did Not Receive Study Product | 5
Safety Analysis Set | 760
Efficacy Analysis Set | 737
Completed | 299
Not Completed | 466
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 9
Not completed — Protocol Violation | 28
Not completed — Lost to Follow-up | 20
Not completed — Death | 377
Not completed — Moved or Changed Medical Team | 23
Not completed — Enrollment in a Clinical Trial | 1
Not completed — Disease Progression | 3
Not completed — Unknown reason | 2

BASELINE CHARACTERISTICS:
Population: Efficacy Analysis Set. Note: 29 participants dd not continue after enrollment.
Arm/Group | Observational Chemotherapy/Bevacizumab
Number analyzed (Participants) | 737
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 347
  >=65 years | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.9)
Gender [Number; unit: participants] — Gender was not recorded for two patients.
  participants
    Female | 293
    Male | 442
Region of Enrollment [Number; unit: participants]
  France | 737

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Kaplan Meier estimates of median progression-free survival according to the metastatic line of treatment, for a median follow-up of 18, 15 and 13 months, respectively
Time Frame: within 36 months
Population: Efficacy analysis set receiving bevacizumab at inclusion
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Bevacizumab With 1st Line Treatment: Patients treated with bevacizumab during first line treatment of chemotherapy
- Bevacizumab With 2nd Line Treatment: Patients treated with bevacizumab during second line treatment of chemotherapy
- Bevacizumab With 3rd Line Treatment: Patients treated with bevacizumab during third line treatment of chemotherapy
Arm/Group | Bevacizumab With 1st Line Treatment | Bevacizumab With 2nd Line Treatment | Bevacizumab With 3rd Line Treatment
Number analyzed (Participants) | 521 | 154 | 62
Months | 10.4 [9.6 to 11.3] | 8.5 [7.0 to 9.2] | 6.3 [4.5 to 8.9]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time between the treatment start (date of the first infusion of bevacizumab) and death from any cause. Kaplan Meier estimates of median overall survival were calculated for the metastatic lines of treatment, with a median follow-up of 18, 15 and 13 months, respectively.
Time Frame: Up to 36 months
Population: Efficacy analysis set receiving bevacizumab at inclusion
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab With 1st Line Treatment | Bevacizumab With 2nd Line Treatment | Bevacizumab With 3rd Line Treatment
Number analyzed (Participants) | 521 | 154 | 62
Months | 25.3 [21.5 to 28.6] | 19.1 [15.7 to 22.6] | 14.9 [11.6 to 20.4]

3. Secondary Outcome: Quality of Life - Global Health Status
Description: Participants rated their quality of life (global health status) on the European Organization for Research and Treatment of Cancer 30-item Core Quality of Life Questionnaire (EORTC QLQ C-30), with total scores ranging from 0 (worst) to 100 (best).
Time Frame: Baseline, 6 and 12 months
Population: Participants in the efficacy analysis set who filled out the questionnaire at inclusion
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Observational Chemotherapy/Bevacizumab
Number analyzed (Participants) | 521
units on a scale
  at Inclusion (n=521) | 67 [50 to 75]
  at Month 6 (n=279) | 67 [50 to 83]
  at Month 12 (n=173) | 67 [50 to 83]
  at Month 18 (n=134) | 67 [50 to 83]

ADVERSE EVENTS:
Time Frame: 36 months
Description: Safety analysis population.
Arm/Group | Observational Chemotherapy/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 74/760
Other Adverse Events (participants affected / at risk) | 353/760
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Chemotherapy/Bevacizumab (N=760)
Embolism Venous (Vascular disorders) | 15 (28)
Embolism (Vascular disorders) | 6 (8)
Hypertension (Vascular disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 13 (15)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 7 (7)
Anal Fistula (Gastrointestinal disorders) | 2 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric Disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1)
Intestinal Fistula (Gastrointestinal disorders) | 1 (1)
Necrotising Colitis (Gastrointestinal disorders) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Impaired healing (General disorders) | 3 (3)
Death (General disorders) | 2 (2)
General Physical Health Deterioration (General disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Urinary Fistula (Renal and urinary disorders) | 1 (1)
Post Procedural Fistula (Injury, poisoning and procedural complications) | 2 (2)
Hepatic Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 3 (3)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Weight Decreased (Investigations) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Anal Haemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Chemotherapy/Bevacizumab (N=760)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 164 (246)
Hypertension (Vascular disorders) | 115 (184)
Embolism venous (Vascular disorders) | 38 (49)
Proteinuria (Renal and urinary disorders) | 118 (215)
Neutropenia (Blood and lymphatic system disorders) | 85 (120)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.